CLINICAL TRIAL: NCT06427135
Title: A Multimodal Wearable Device-based Study to Evaluate the Efficacy of an Exercise Prescription Intervention in Inflammatory Bowel Disease: a Single-center, Randomized Controlled Trial
Brief Title: A Multimodal Wearable Device-based Study to Evaluate the Efficacy of an Exercise Prescription Intervention in IBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ping An (Other)
Responsible Party: Sponsor-Investigator, Ping An, Professor, Renmin Hospital of Wuhan University
Organization: Renmin Hospital of Wuhan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2024-K058
Record Dates: First submitted 2024-04-25; First posted 2024-05-23 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Exercise interventions; Inflammatory Bowel Diseases; Wearable Device
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized controlled study divided into intervention and control groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise interventions (Experimental): Adding exercise intervention therapy to existing medications
  Interventions: Behavioral: Exercise interventions
- Conventional drug therapy (No Intervention): No exercise intervention, use of existing medication.

INTERVENTIONS:
Behavioral: Exercise interventions — Rehabilitation physician or rehabilitation therapist, to engage in physical exercise or patients, according to the medical examination data (including exercise test and physical strength test), according to their health, physical strength, and cardiovascular function status, with the form of a prescription for the type of exercise, intensity of exercise, exercise time and frequency of exercise, to put forward the precautions to be taken during exercise.
  Arms: Exercise interventions

SUMMARY:
This project is a multimodal wearable device-based evaluation of the efficacy of an exercise prescription intervention for inflammatory bowel disease in a This is a single-center, randomized controlled clinical study to evaluate the efficacy of an exercise prescription intervention in inflammatory bowel disease based on multimodal wearable devices. The experimental group was treated with exercise intervention therapy on top of the existing medication.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic inflammatory bowel disease that mainly involves the digestive system, including Crohn's disease (CD) and ulcerative colitis (UC).CD is characterized by abdominal pain, diarrhea, abdominal mass, fistula formation and intestinal obstruction. CD is characterized by abdominal pain, diarrhea, abdominal mass, fistula formation, and intestinal obstruction; UC is characterized by diarrhea, mucopurulent blood stools, and abdominal pain, and the peak age of onset is between 15 and 40 years old. Notably, many studies have shown that patients with inflammatory bowel disease commonly suffer from malnutrition, low body mass index (BMI), muscle atrophy, decreased bone density, and fatigue and anxiety, and that surgery is not a one-time event, with patients often requiring several surgeries.

Current treatment strategies focus on medication, nutritional support and nursing care, neglecting other possible adjunctive treatments.

Exercise interventions, as an effective adjunctive therapy for inflammatory bowel disease, have been shown to have anti-inflammatory, anti-muscle atrophic, and physical enhancement effects, improve psychological status, and also have beneficial effects on intestinal flora and intestinal absorption. Exercise is also economical, efficient and highly feasible, making it more acceptable to IBD patients. With the integration of physical medicine and the implementation of Healthy China, the role of exercise intervention in the majority of patients will be more important and its application will be more extensive.

Multimodal wearable device is a simple and efficient miniaturized smart device commonly used in the field of exercise, which can monitor the wearer's heart rate, blood oxygen, step count, exercise data in real time, etc. This group proposes to combine the multimodal wearable device as an auxiliary device with the exercise intervention for patients with inflammatory bowel disease (IBD), which is the first of its kind in China.

Most of the current studies are conducted on the conditions of small samples, single period, and single exercise modality, lack of studies on large samples and multi index evaluation, and the field has not yet formed a unified consensus on personalized exercise intervention for different levels of patients. There is still considerable work to be done on the study of exercise interventions for the treatment of inflammatory bowel disease.

Therefore, this group proposes to conduct a randomized controlled trial to investigate the effects of exercise intervention on body composition and disease progression in patients with inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Commitment to comply with the study procedures and cooperate in the implementation of the full study
* Age ≥ 18 years old, gender is not limited
* Muscle strength examination of all four limbs is greater than or equal to grade 3
* Patients with a diagnosis of CD or UC in combination with clinical presentation, laboratory examination, endoscopy, imaging and histopathologic examination, with a disease course in mild to moderate activity or remission
* Presence of low or high BMI, malnutrition, muscular dystrophy, and anxiety
* Voluntarily sign a written informed consent

Exclusion Criteria:

* Absolute contraindications to exercise: acute stages of various diseases (e.g. cerebral hemorrhage, acute stage of myocardial infarction), severe complications, severe cardiopulmonary dysfunction, severe gastrointestinal problems (e.g. gastric perforation, intestinal obstruction), severe locomotor system disorders (e.g. severe bone fracture), as well as other diseases that are not under effective control
* Relative contraindications to exercise: severe hypertension, severe diabetes, chronic pain, cardiac arrhythmia, etc
* Persons with unstable vital signs
* Presence of cognitive, communication disorders
* Patients who have recently undergone gastrointestinal surgery (<1 month) or who have not fully healed
* Short bowel syndrome
* Presence of extra-intestinal manifestations and complications that interfere with therapy, such as retinopathy, deep vein thrombosis, etc
* Pregnant or lactating women
* Active tuberculosis; if subjects are suspected of having active tuberculosis, chest X-ray, sputum and exclusion by clinical signs and symptoms are required
* Other potential subjects who are not suitable for participation in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
skeletal muscle mass index | Weeks 0, 4, 8, 12 and 16 of treatment
  Changes in skeletal muscle mass index (SMI) were detected using a body composition analyzer, and were considered statistically significant if they were higher in the intervention group than in the control group (P < 0.05);Skeletal muscle mass index is calculated as the ratio of limb skeletal muscle mass (kg) to height (m) in kg/m^2.

SECONDARY OUTCOMES:
Quality of life rating | Weeks 0, 4, 8, 12 and 16 of treatment
  Changes before and after the intervention were assessed by means of a quality of life questionnaire (Inflammatory Bowel Disease Questionnaire, IBDQ) with a total score of 224, the higher the better.
Psychological assessment | Weeks 0, 4, 8, 12 and 16 of treatment
  Changes before and after the intervention were assessed by means of the Anxiety and Depression Scale (Hospital Anxiety and Depression Scale, HADS), with a total HADS score of 42, with higher scores indicating worse indicators.
Fatigue status assessment | Weeks 0, 4, 8, 12 and 16 of treatment
  Changes before and after the intervention were assessed by means of a fatigue scale (Functional Assessment of Chronic Illness Therapy, FACIT), with a total FACIT score of 52, with a higher score indicating a better indicator.
body fat percentage | Weeks 0, 4, 8, 12 and 16 of treatment
  Detecting changes in subjects' body fat percentage using a body composition analyzer
muscle power | Weeks 0, 4, 8, 12 and 16 of treatment
  Changes in muscle strength (kg) in the limbs of the subjects were detected using a plyometer.
spirometry | Weeks 0, 4, 8, 12 and 16 of treatment
  Changes in spirometry (mL) before and after the intervention were tested using an electronic spirometry tester.
Fecal calprotectin level | Weeks 0, 4, 8, 12 and 16 of treatment
  Test for changes in fecal calprotectin (FCP) levels in subjects before and after the intervention.The normal range for FCP is less than 100 ng/mL.
C-reaction protein level | Weeks 0, 4, 8, 12 and 16 of treatment
  To test for changes in subjects' C-reactive protein (CPR) levels before and after the intervention.The normal range for CRP is less than 5.2 mg/l for adult males and less than 4.6 mg/l for adult females.

CONTACTS AND LOCATIONS:
Overall Officials: Ping An, Principal Investigator — Renmin Hospital of Wuhan University

IPD SHARING:
Plan to Share IPD: No